CLINICAL TRIAL: NCT02043288
Title: A Phase III, Open-label, Randomized Study of the Combination Therapy With NC-6004 and Gemcitabine Versus Gemcitabine Alone in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Combination Therapy With NC-6004 and Gemcitabine Versus Gemcitabine Alone in Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orient Europharma Co., Ltd. (Industry)
Collaborators: NanoCarrier Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NC-6004-005
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic cancer; Platinum; Micelle
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — demplatin pegraglumer; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NC-6004 and Gemcitabine combination (Experimental): NC-6004 90mg/m2 i.v. on Day 1 and Gemcitabine 1000mg/m2 i.v. on Day 1 and Day 8 respectively
  Interventions: Drug: NC-6004; Drug: Gemcitabine
- Gemcitabine monotherapy (Active Comparator): Gemcitabine 1000mg/m2 i.v. on Day 1 ,8 and 15
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: NC-6004 — Study group (3 week/cycle):
  NC-6004 90 mg/m2 i.v. inf. over 60 min on Day 1
  Other Names: Micelplatin
  Arms: NC-6004 and Gemcitabine combination
Drug: Gemcitabine — Study group (3 week/cycle):
  Gemcitabine 1000 mg/m2 i.v. inf. over 30 min on Day 1 and Day 8 (follow by administration of NC-6004)
  Control group (4 week/cycle):
  Gemcitabine 1000 mg/m2 i.v. inf. over 30 min on Day 1, Day 8 and Day 15
  Other Names: Gemzar

SUMMARY:
This clinical trial is designed to evaluate the impact of the addition of NC-6004 to gemcitabine in the treatment of patients with locally advanced or metastatic pancreatic cancer in Asian countries.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the most deadly cancers because of the predominately late diagnosis. Gemcitabine (GEM) is the standard treatment for advanced and metastatic pancreatic cancer. According to preclinical data and few early phase studies, a combined use of gemcitabine and cisplatin (CDDP) showed synergistic efficacy against pancreatic cancer. NC-6004, a novel micellar cisplatin formulation, retains the activity but avoids the renal toxicity and neurotoxicity caused by the high peak Cmax concentrations of cisplatin. This trial is designed to evaluate the impact of the addition of NC-6004 to gemcitabine in the treatment of patients with locally advanced or metastatic pancreatic cancer.

The main hypothesis of this study is that NC-6004 plus gemcitabine combination is superior to gemcitabine alone in terms of overall survival in locally advanced or metastatic pancreatic cancer patients

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged between 20 to 80 years (inclusive)
2. Unresectable, histologically or cytologically confirmed, locally advanced or metastatic pancreatic cancer (adenocarcinoma, adenosquamous carcinoma or poorly differentiated carcinoma)
3. Presence of at least one measurable tumor lesion (longest diameter ≥ 10 mm)
4. No prior systemic anti-cancer therapy* and radiotherapy** for advanced pancreatic cancer

   * Patients with post-operative adjuvant chemotherapy other than platinum products (e.g. cisplatin, carboplatin and oxaliplatin, etc.) or radiotherapy or chemo-radiotherapy completed more than 6 months before recurrence will be eligible.

   ** Patients with prior palliative radiotherapy of < 20% bone marrow involvement prior to 6 months from screening will be eligible.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
6. Adequate organ function defined as:

   * 3,000 cells/μL ≤ WBC ≤ 12,000 cells/μL
   * Absolute neutrophils count (ANC) ≥ 1,500 cells/μL
   * Platelets ≥ 100,000 cells/μL
   * Hemoglobin (Hb) ≥ 9.0 g/dL
   * Alanine amino transferase (ALT) and aspartate amino transferase (AST) ≤ 2.5 times the upper limit of normal (ULN) in patients with no demonstrable hepatic metastasis, or ≤ 5 x ULN in patients with hepatic metastasis
   * Serum bilirubin ≤ 1.5 x ULN in patients with no demonstrable hepatic metastasis and obstructive jaundice, or ≤ 2.5 x ULN in patients with hepatic metastasis or obstructive jaundice
   * Serum creatinine (SCr) ≤ 1.5 mg/dL and creatinine clearance (CrCl) ≥ 60 mL/min (from 24-hour urine test or Cockcroft-Gault formula)
   * Corrected serum calcium ≤ ULN
7. If fertile*, willing to use barrier contraception till 6 months after the end of treatment

   * With the following exceptions: 1) pre-menopausal females with bilateral tubal ligation, bilateral oophorectomy or hysterectomy; 2) post-menopausal women, defined as 12 months of spontaneous amenorrhea; 3) males with vasectomy.
8. Willing and able to comply with study procedures and provide written informed consent

Exclusion criteria:

1. Pregnancy or breastfeeding
2. Active concomitant malignancy or history of other cancer except carcinoma in situ of cervical squamous cell carcinoma, stage I colon cancer or other malignance that has remained disease-free for more than 3 years after curative intervention
3. Metastasis to the central nervous system or brain
4. Evidence of hearing impaired ≥ Grade 2 as assessed by pure tone audiometry or other neurotoxicity ≥ Grade 2

   * Patients with age-associated hearing loss at the high frequencies that, in the judgment of the investigator, would not interfere significantly with patient's safety or study assessments will be eligible to enroll.
5. Patient with pulmonary fibrosis or interstitial pneumonia
6. Marked pleural effusion or ascites above Grade 2
7. Patient with known HIV infection
8. Patient with active hepatitis B, hepatitis C or any other ongoing severe infections
9. Patient with severe mental disorder
10. As judged by the investigator, any evidence of significant laboratory findings or severe/uncontrolled clinical disorders (e.g. dementia, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, unstable angina, active cardiomyopathy, unstable arrhythmia, and other unstable or uncompensated respiratory, cardiac, hepatic, renal and/or infectious disease)
11. Patient with known hypersensitivity to Pt compounds
12. Known severe drug hypersensitivity
13. Treatment with a non-approved or investigational product within 30 days before Day 1 of study treatment
14. Alcoholic liver disease* or liver disease with obvious clinical symptom or sign

    * the investigator should judge from medical examination by interview and laboratory test including γ-GTP, AST and ALT
15. Daily Alcohol consumption within 6 months before the screening as an average weekly intake of >21 units (168 g of pure alcohol) or an average daily intake of >3 units (24 g of pure alcohol) for males / an average weekly intake of >14 units (112 g of pure alcohol) or an average daily intake of >2 units (16 g of pure alcohol) for females.

    Kind of Alcohol Alcohol Percentage mL per 1 unit =8 g of pure alcohol

    Beer 5 % 200 mL

    Whiskey/Brandy 40 % 25 mL

    Wine 12 % approx. 83 mL

    Sake 15 % approx. 67 mL

    Distilled spirit 25 % 40 mL

    Kaoliang 50 % 20 mL
16. Patient with uncontrolled diabetes
17. Radiotherapy within 6 months before screening
18. Experienced Abdominal Radiotherapy
19. Experienced treatment of Gemtuzumab ozogamicin
20. Patient with autoimmune hepatitis or idiopathic thrombocytopenic purpura (ITP)
21. Observation of "attenuated or reversed hepatic venous portal blood flow*" was confirmed by doppler ultrasonography or CT (recommend evaluation in arterial phase, portal-venous phase and equilibrium phase) of the liver * On doppler ultrasonography of right and left branch of portal vein, blood flow is measured as about 0 mL/min or between plus and minus, which indicate obvious blood flow obstruction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 3.5 years
  Overall survival is defined as the time from the treatment initiation until death from any cause, and censored at the last follow up time.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 3.5 years
  Progression free survival is defined as the time from the treatment initiation until progression or death, and censored at the last follow up time.
Response rate (RR) and disease control rate (DCR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria | 3.5 years
  * Response rate is defined as counts and proportions of patients responding complete response or partial response within the duration of the study.
  * Disease control rate is defined as counts and proportions of patients responding complete response, partial response or progressive disease within the duration of the study.
Duration of response | 3.5 years
  * Duration of overall response (DOR) will be measured from the time of initial response (CR or PR) until documented progression or death, and censored at last follow up time.
  * Duration of stable disease (DSD) will be measured from the time of initial stable disease (SD) until documented progression or death, and censored at last follow up time.
CA19-9 | 3.5 years
  CA19-9 values and changes from baseline will be summarized.
Quality of life (QoL) using EORTC QLQ-C30 | 3.5 years
  Quality of life (QoL) values and changes from baseline will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D., Ph. D., Principal Investigator — National Institute of Cancer Research, National Health Research Institutes
Locations (43):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Japan (16):
  - Aichi Cancer Center, Aichi
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - Saitama Cancer Center, Saitama
  - National Hospital Organization Shikoku Cancer Center, Shikokuchūō
  - Shizuoka Cancer Center, Shizuoka
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - Kyorin university Hospital, Tokyo
  - National Cancer Center Hospital East, Tokyo
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Malaysia (2):
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
- Makati Medical Center, Makati, Philippines
- National Cancer Centre, Singapore, Singapore
- South Korea (5):
  - Ajou University Hospital (AUH), Gyeonggi-do
  - Samsung Medical Center (SMC), Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital (CUK SSMH), Seoul
  - Korea University Guro Hospital (KUGH), Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
- Taiwan (16):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University-Shuang-Ho Hospital, Ministry of Health and Welfare, Taipei
  - Chang Gung Memorial Hospital, Linkou Branch, Taipei
  - Chi Mei Medical Center, Yongkang District

IPD SHARING:
Plan to Share IPD: No